CLINICAL TRIAL: NCT06702852
Title: Investigation of the Predictive Value of Near Infrared Spectroscopy in Chronic Lower Extremity and Other Chronic Non-healing Ulcers
Brief Title: Effect of NIRS-assisted Assessment on Chronic Lower Extremity and Other Chronic Non-healing Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to significant protocol deviations in the execution of the study that compromised data integrity. These deviations were unrelated to the safety or performance of the investigational device.
Sponsor: Kent Imaging Inc (Industry)
Collaborators: WoundCentrics LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MG-NIRS-03
Record Dates: First submitted 2024-10-03; First posted 2024-11-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Ulcers
Keywords: tissue oxygenation; Near infrared spectroscopy; lower extremity ulcers; ulcers; SnapshotNIR; NIRS; imaging; oxyhemoglobin; deoxyhemoglobin; hemoglobin; oxygen saturation; wound healing
MeSH Terms: conditions — Ulcer; Leg Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): The control group will receive the standard of care per the facility Standard Operating Procedures (SOP)
- Intervention (Experimental): The intervention group will receive the standard of care per the facility Standard Operating Procedures (SOP) with the addition of NIRS imaging utilizing the SnapshotNIR
  Interventions: Device: NIRS imaging in addition to SOC

INTERVENTIONS:
Device: NIRS imaging in addition to SOC — The intervention group will receive the standard of care per the facility Standard Operating Procedures (SOP) with the addition of NIRS imaging utilizing the SnapshotNIR
  Arms: Intervention

SUMMARY:
Investigation of the predictive value of Near Infrared Spectroscopy in Chronic Lower Extremity and Other Chronic non-healing Ulcers

DETAILED DESCRIPTION:
The objective of this study is to evaluate the clinical and economical effect of introduction of near-infrared spectroscopy (NIRS) in the diagnostic and treatment protocol of patients with lower extremity (LE) ulcers as well as other chronic non-healing ulcers, and to determine a positive and/or negative predictive value or range of values for NIRS correlating to patient progress and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current patients or patients admitted to Christus Wound Care and Hyperbaric Medicine Departments between July 1, 2024, and December 31, 2024, for the treatment of lower extremity ulcers and other chronic non-healing ulcers.
* Lower extremity ulcers and chronic non-healing ulcers will be included in the study regardless of the wound/ulcer etiology. Patients may become eligible for the study at any point during their course of treatment.

Exclusion Criteria:

* Patients who are being treated at multiple research sites simultaneously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Patient health outcome | From enrollment to closeout or 12 weeks from enrollment whichever is earlier
  To evaluate the impact of the addition of NIRS to the SOP on patient health outcome by comparing between the control and interventional groups

SECONDARY OUTCOMES:
Health Economic Impact | From enrollment to closeout or 12 weeks from enrollment whichever is earlier
  To evaluate the impact of the addition of NIRS to the SOP on treatment plans, interventions, and financial expenses by comparing between the control and interventional groups

CONTACTS AND LOCATIONS:
Overall Officials: Marcus L Gitterle, MD, Principal Investigator — CHRISTUS Santa Rosa Hospital Wound Care and Hyperbaric Center - San Antonio, Westover Hills, San Marcos and New Braunfels
Locations (3):
- United States (3):
  - Christus Santa Rosa Wound Care and Hyperbaric Center, New Braunfels, Texas
  - Christus Santa Rosa Wound Care and Hyperbaric Center, San Antonio, Texas
  - Christus Santa Rosa Wound Care and Hyperbaric Center, San Marcos, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serena TE, Yaakov R, Serena L, Mayhugh T, Harrell K. Comparing near infrared spectroscopy and transcutaneous oxygen measurement in hard-to-heal wounds: a pilot study. J Wound Care. 2020 Jun 1;29(Sup6):S4-S9. doi: 10.12968/jowc.2020.29.Sup6.S4. PMID 32530756
- [Background] Geskin G, Mulock MD, Tomko NL, Dasta A, Gopalakrishnan S. Effects of Lower Limb Revascularization on the Microcirculation of the Foot: A Retrospective Cohort Study. Diagnostics (Basel). 2022 May 26;12(6):1320. doi: 10.3390/diagnostics12061320. PMID 35741130
- [Background] Farber A. Chronic Limb-Threatening Ischemia. N Engl J Med. 2018 Jul 12;379(2):171-180. doi: 10.1056/NEJMcp1709326. No abstract available. PMID 29996085
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in diabetes since 1980: a pooled analysis of 751 population-based studies with 4.4 million participants. Lancet. 2016 Apr 9;387(10027):1513-1530. doi: 10.1016/S0140-6736(16)00618-8. Epub 2016 Apr 6. PMID 27061677